CLINICAL TRIAL: NCT07003724
Title: Patients' Awareness, Attitude and Trust in the Use of Artificial Intelligence in Dentistry
Brief Title: Patient's Knowledge About AI in Dentistry
Status: Not yet recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Merna Ezzat Boules Malek, DOCTOR, Cairo University
Other Study IDs: 566889877890
Record Dates: First submitted 2025-05-26; First posted 2025-06-04 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-05

CONDITIONS: Patients Attitude on AI in Dentistry; Trust AI; Concerns on AI
Keywords: Artificial intelligence in dentistry

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients at Public Hospitals and Universities hospitals: Patients seeking dental treatment at Public Hospitals and University Hospitals
  Interventions: Other: Questionaire
- Patients at Private Clinics: Patients seeking dental treatments at Private Clinics
  Interventions: Other: Questionaire

INTERVENTIONS:
Other: Questionaire — Questionnaire evaluating level of awareness of patients towards using AI in dentistry

SUMMARY:
It's a cross sectional study , A validated questionnaire to knows patients attitude , opinion towards using AI in dentistry used before By Ayad et al on a different population.

DETAILED DESCRIPTION:
The purpose of this study is to investigate public awareness, perceptions and attitudes about the application of AI in dentistry and also patients' worries as many ethical concerns may be in people's mind as algorithim unfairness, data privacy, and the possibility of employment displacement in the dental industry, by distributing a survey to a wide range of dental patients from public hospitals and private clinics , this study aims to know patient's opinions regarding the possible advantages , disadvantages , ethical concerns , and patients thoughts on using AI .

ELIGIBILITY:
Inclusion Criteria:

* Age range between 25 to 50
* Females and males
* Low, middle and high socioeconomic
* Egyptian patients
* acceptable educational level
* patients in dental waiting areas

Exclusion Criteria:

* Anyone above or below the age range mentioned (25-50 years )
* Special needs patients
* Non-Egyptian patients
* Non-Educated patients
* very low socio-economic class
* patients in other waiting areas rather than dental ones

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients seeking dental treatment either in Public Hospitals, Universities hospitals ,or Patients in Private dental clinics
Sampling Method: Probability Sample
Enrollment: 382 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of Public Awareness via Questionnaire | 6 Months
  Quantify the level of public awareness about AI and its potential applications in dentistry via Questionnaire to assess outcome measure

SECONDARY OUTCOMES:
Evaluation of Public Perception Via Questionnaire | 6 Months
  Determine public attitudes towards AI-powered dental technologies, including perceived benefits and risks through questionnaire to assess outcome measure

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided